CLINICAL TRIAL: NCT06985940
Title: Visual and Acoustic Effects of Human Thermal Comfort and Perception in a Micro-Climatically Steady Environment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lab schedule, Resources
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-1656; A489400 (Other: UW Madison); L&S/PLANNING & LANDSCAPE ARCH (Other: UW Madison)
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Thermal Perception
MeSH Terms: interventions — Photic Stimulation; Acoustic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Climate-controlled chamber (Experimental): Participants will be in a climate-controlled chamber. Temperature will vary by 5 degrees both warmer and colder.
  Interventions: Other: Visual stimulation; Other: Acoustic stimulation; Other: Combination

INTERVENTIONS:
Other: Visual stimulation — Participants will watch a 10-minute snow- or fire-themed video
Other: Acoustic stimulation — Participants will listen to a natural sound from fire burning or snow falling
Other: Combination — Participants will undergo both visual and acoustic stimulation

SUMMARY:
The goal of this clinical trial is to understand how environmental factors influence comfort and health. The main question it aims to answer is:

* do temperature, visuals, and sounds affect a person's physiology and perception?

Participants will watch short videos in 2 different climate-controlled environments and provide feedback on their thermal experiences.

DETAILED DESCRIPTION:
Participants will engage in a series of sessions in a climate-controlled environment, where researchers will manipulate temperature, visuals, and sounds to study their effects on various physiological measurements, including blood pressure, pulse rate, core temperature, and skin temperature. The study will take place in two distinct chambers, with each chamber designed to allow for precise control of environmental variables. Participants will be asked to watch short video clips in different thermal environments and provide feedback on their thermal experiences.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* BMI between 18-27.5 kg/m²
* No history of color blindness or sensory impairments
* Normal chronotype (consistent sleep-wake patterns)
* Must have lived in or near Guangzhou, China for at least two months prior to participation

Exclusion Criteria:

* Children (age under 18), elders (age > 60)
* People with obesity
* People with a history of color blindness
* People without a consistent sleep-awake pattern
* People with limited English proficiency

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in thermal perception | Baseline to 90 minutes
  Thermal comfort will be assessed using a visual analogue scale (VAS) to measure perceptions of thermal sensation, preference, comfort, pleasantness, and self-perceived shivering. The thermal acceptance of the environment will be rated on a binary scale (acceptable/unacceptable).
Change in pulse rate | Baseline to 90 minutes
  Pulse will be measured using the Empatica Plus 4
Change in skin temperature | Baseline to 90 minutes
  Skin temperature will be measured at 14 sites using iButtons (DS1922L)
Change in blood pressure | Baseline to 90 minutes
  Measured using an automatic blood pressure monitor
Change in core temperature | Baseline to 90 minutes
  Measured using CORE core temperature device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes